CLINICAL TRIAL: NCT00996008
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Multi-Centre Study of the Safety and Efficacy of CT 327, Pegylated K-252, Formulated as a Cream, When Administered Twice Daily for 14 Days to Subjects With Mild-to-Moderate Atopic Dermatitis
Brief Title: CT 327 in the Treatment of Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow recruitment, study was stopped before target enrollment was achieved
Sponsor: Creabilis SA (Industry)
Responsible Party: Professor Peter Itin, University Hospital, Basel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT 327 AD 02-09
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Mild to Moderate Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo only (Placebo Comparator): Subjects will apply placebo cream to all 4 target lesions
  Interventions: Drug: placebo
- Active plus placebo (Active Comparator): Subjects will receive CT 327 on 2 of 4 target lesions located on one side of their body. On the remaining 2 target lesions on the other side of their body, placebo will be applied.
  Interventions: Drug: CT 327

INTERVENTIONS:
Drug: placebo — 0.5 g (w/w) placebo cream applied to each target lesion twice daily
  Arms: Placebo only
Drug: CT 327 — 0.5 g CT 327 cream will be applied to 2 target lesions twice daily 0.5 g placebo cream will be applied to remaining 2 target lesions twice daily
  Arms: Active plus placebo

SUMMARY:
This study will look at how safe and effective, a novel agent, CT 327 cream is in treating patients with mild to moderate atopic dermatitis (AD). Patients will be treated twice daily for 14 days on specific lesions of AD and safety and symptoms of AD will be assessed throughout the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects aged >18 year
* Written informed consent
* Mild to moderate AD at baseline (EASI score of at least 2 or 3)
* Active AD (visible eczema, erythema and pruritus)
* Presence of at least four target lesions (symmetrically) at inclusion (ideally at the elbow flexions and knee bends)

Exclusion Criteria:

* If female of childbearing potential not using an adequate and appropriate form of contraception such as oral contraceptive; intra-uterine device (IUD); contraceptive injection, implant or patch
* If female, are pregnant or lactating, or intend to become pregnant during the study period
* Allergy to test drug or excipients
* Usage of topical corticosteroids or other topical treatments for AD within the last two weeks prior to study entry (including calcineurin inhibitor, topical H1 and H2 antihistamines, topical antimicrobials, other medicated topical agents) or herbal preparation to the area selected for treatment
* Within 4 weeks prior to study entry, have received systemic treatment for atopic dermatitis (including systemic corticosteroids, nonsteroidals, immunosuppressants, or immunomodulating drugs, or treatment with light).
* Presence of major medical illness requiring systemic therapy including cancers
* Clinical diagnosis of bacterial infection of the skin including impetigo and abscesses
* Any clinical relevant ECG abnormality
* Have any clinically significant abnormal clinical laboratory test results at screening
* Received any investigational drug or taking part in any clinical study within three months prior to this study
* History of drug, alcohol or other substance abuse or other factors limiting the ability to co-operate and to comply with this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of CT 327 vs Placebo in terms of improvements from baseline on Modified Eczema Area Severity Index (mEASI) score: Proportion of subjects with a reduction in mEASI-score of ≥ 50% on day 14 | 14 days

SECONDARY OUTCOMES:
To assess the efficacy of a 14-days treatment of CT 327 vs Placebo in terms of improvements from baseline on: Proportion of subjects with a reduction in m-EASI-score of > 75% on day 14 | 14 days

CONTACTS AND LOCATIONS:
Locations (5):
- Switzerland (5):
  - University Hospital, Basel
  - Inselspital, Bern
  - CHUV, Hôpital de Beaumont, Lausanne
  - Kantonsspital St Gallen, Sankt Gallen
  - University Hospital, Zurich